CLINICAL TRIAL: NCT03523117
Title: A Multicenter, Randomized, Active-Controlled Study to Investigate the Efficacy and Safety of Intravenous Ferric Carboxymaltose in Pediatric Patients With Iron Deficiency Anemia
Brief Title: Multicenter Randomized Active-controlled Study to Investigate Efficacy & Safety of IV FCM in Pediatric Patients With IDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT17044
Record Dates: First submitted 2018-04-17; First posted 2018-05-14 (Actual); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; ferrous sulfate; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferric Caroboxymaltose (Active Comparator): Ferric Carboxymaltose - 2 doses (day 0 and day 7) at 15 mg/kg to a maximum single dose of 750 mg (whichever is smaller) up to a maximum of total dose of 1500 mg administered as either an undiluted IV push at a rate of 100 mg (2mL)/minute OR in no more than 250 mL of normal saline and infused over 15 minutes.
  Interventions: Drug: Ferric carboxymaltose
- Oral Ferrous Sulfate (Active Comparator): Oral Ferrous Sulfate - will receive an age-dependent formulation of oral ferrous sulfate daily for 28 days as follows: participants <12 years of age will receive 6 mg (elemental iron)/kg/day divided into 2 daily doses of an oral liquid formulation, either drops or elixir, and participants ≥12 will receive 2 daily doses of oral tablets. Infants and children (ages 1 to <4 years) will receive oral ferrous sulfate drops, while children (ages ≥4 to <12 years) will receive oral ferrous sulfate elixir. Adolescents (ages ≥12 to 17 years) will receive an oral ferrous sulfate tablet (65 mg of elemental iron/tablet/dose) twice a day (BID). The maximum daily dose for all participants is 130 mg of elemental iron.
  Interventions: Drug: Ferrous Sulfate

INTERVENTIONS:
Drug: Ferric carboxymaltose — Intravenous iron
  Other Names: Injectafer; Ferinject
  Arms: Ferric Caroboxymaltose
Drug: Ferrous Sulfate — oral iron therapy
  Other Names: oral iron
  Arms: Oral Ferrous Sulfate

SUMMARY:
The primary objective of this study is to demonstrate the efficacy and safety of intravenous ferric carboxymaltose (FCM), compared to oral iron, in pediatric participants who have iron deficiency anemia.

DETAILED DESCRIPTION:
This is a Phase III, multicenter, randomized, active-controlled study that compares the efficacy and safety of FCM to oral iron in pediatric participants with IDA and a documented history of an inadequate response to oral iron therapy at least 8 weeks (56 days) prior to randomization.

Participants who satisfy the inclusion requirements and no exclusion criteria will be eligible to participate in this study and enter into a screening phase to confirm eligibility. Randomization will occur via the Interactive Response Technology (IRT) system in a 1:1 ratio to either Group A, participants receiving FCM, or Group B, participants receiving oral iron (oral solution drops, elixir or oral tablets). Randomization will be stratified by baseline Hgb (<10, ≥10 g/dL) and age (1 to <12 years and ≥12 to 17 years).

The oral ferrous sulfate formulation received will be based on the participant's age, such that infants and children (1 to <4 years of age) will receive ferrous sulfate drops, children (≥4 to <12 years of age) will receive ferrous sulfate elixir, and adolescents (≥12 to 17 years of age) will receive ferrous sulfate tablets. Participants who experience adverse clinical symptoms due to the oral iron during the treatment phase may have a weight-based dose of ferrous sulfate reduced from 6 mg/kg to 3 mg/kg. If the participant is receiving tablets, the dose will be reduced from one tablet taken twice daily to one tablet per day.

Once randomized, all participants will return for efficacy and safety evaluations, including adverse events and laboratory assessments, on Days 7, 14, 28, and 35. Additional pharmacokinetic sampling and analyses will be performed for participants receiving FCM on Days 0 and 7.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 1 to 17 years of age with assent to participation and his/her parent or guardian is willing and able to sign the informed consent approved by the Independent Review Board / Ethics Committee.
2. Screening Hgb <11 g/dL.
3. Screening ferritin ≤300 ng/mL and transferrin saturation (TSAT) <30%.
4. Participants must have a documented history of an inadequate response to any oral iron therapy for at least 8 weeks (56 days) prior to randomization.
5. For participants who are receiving an erythropoietin stimulating agent (ESA): stable ESA therapy (+/- 20% of current dose) for at least 8 weeks prior to the qualifying screening visit and no ESA dosing or product changes anticipated for the length of the trial.
6. Participants undergoing treatment for inflammatory bowel disease (IBD) must be on stable therapy for at least 8 weeks prior to consent.

Exclusion Criteria:

1. Known history of hypersensitivity reaction to any component of FCM.
2. Previous randomization and treatment in this study or any other clinical study of FCM or VIT-45.
3. History of acquired iron overload, hemochromatosis, or other iron accumulation disorders.
4. Chronic kidney disease participants on hemodialysis.
5. History of significant diseases of the liver, hematopoietic system, cardiovascular system, psychiatric disorder, or other conditions which, on the opinion of the investigator, may place a subject at added risk for participation in the study.
6. Any existing non-viral infection.
7. Known history of positive hepatitis B antigen (HBsAg) or hepatitis C viral antibody (HCV) with evidence of active hepatitis.
8. Known history of positive HIV-1/HIV-2 antibodies (anti-HIV).
9. Anemia due to reasons other than iron deficiency (e.g., hemoglobinopathy and vitamin B12 or folic acid deficiency) that has not been corrected.
10. Intravenous iron and /or blood transfusion in the 4 weeks prior to consent.
11. Administration and / or use of an investigational product (drug or device) within 30 days of screening.
12. Alcohol or drug abuse within the past six months.
13. Female participant who is pregnant or lactating, or sexually active female who are of childbearing potential not willing to use an acceptable form of contraceptive precautions during the study.
14. Unable to comply with study procedures and assessments

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Falone, Study Director — American Regent, Inc.
Locations (16):
- United States (16):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - International Research Partners, Inc., Doral, Florida
  - ProHealth Research Center, Doral, Florida
  - Garden Medical Research, Inc., Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida
  - Riley Hospital for Children,Room 4340, Indianapolis, Indiana
  - Caro Health Plaza, Caro, Michigan
  - Galen Research, Chesterfield, Missouri
  - Tiga Pediatrics, PC, The Bronx, New York
  - Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Texas Children Hospital, Houston, Texas
  - Tekton Research, San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 3, multicenter, multinational, randomized, active-controlled study that compared the efficacy and safety of FCM to oral iron in pediatric participants with IDA and a documented history of an inadequate response to oral iron at least 8 weeks (56 days) prior to randomization.
  Participants who satisfied the inclusion requirements and no exclusionary criteria were eligible to participate in this study and enter into a screening phase to confirm eligibility.
Period: Overall Study
Arm/Group | Ferric Caroboxymaltose | Oral Ferrous Sulfate
Started | 40 | 39
Completed | 39 | 37
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Caroboxymaltose | Oral Ferrous Sulfate | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Customized [Mean (Standard Deviation); unit: years] | 12.5 (.5) | 12.8 (.4) | 12.6 (.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin g/dL
Description: Change in hemoglobin g/dL from baseline to day 35 will be analyzed using parametric analysis of covariance (ANCOVA). The model will include terms for the randomization strata (hemoglobin and age categories), baseline hemoglobin, as well as treatment group. Baseline hemoglobin will be defined as the last hemoglobin obtained before randomization.
Time Frame: Baseline to day 35
Population: Intent to Treat (ITT)
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Ferric Caroboxymaltose | Oral Ferrous Sulfate
Number analyzed (Participants) | 40 | 39
g/dL | 2.22 [1.69 to 2.75] | 1.92 [1.43 to 2.41]
Statistical Analysis 1: Comparison: Ferric Caroboxymaltose vs Oral Ferrous Sulfate; Test type: Superiority; p = 0.3108, ANCOVA; Mean Difference (Final Values) = 0.30

2. Secondary Outcome: Change in Ferritin µg/L From Baseline to Day 35
Description: Change in ferritin µg/L from baseline to day 35 was analyzed using parametric analysis of covariance (ANCOVA). The model included terms for the randomization strata (hemoglobin and age categories), baseline ferritin as a covariate.
Time Frame: Baseline to day 35
Population: intent to treat (ITT) all randomized
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/L
Arm/Group | Ferric Caroboxymaltose | Oral Ferrous Sulfate
Number analyzed (Participants) | 40 | 39
µg/L | 2.22 [1.69 to 2.75] | 1.92 [1.43 to 2.41]
Statistical Analysis 1: Comparison: Ferric Caroboxymaltose vs Oral Ferrous Sulfate; Test type: Superiority; p = 0.0001, ANCOVA; Mean Difference (Final Values) = 0.30

3. Secondary Outcome: Change in TSAT (%) From Baseline to Day 35
Description: Change in TSAT (%) from baseline to day 35 was analyzed using parametric analysis of covariance (ANCOVA). The model included terms for the randomization strata (hemoglobin and age categories), baseline ferritin as a covariate
Time Frame: Baseline to day 35
Population: Intent to treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | Ferric Caroboxymaltose | Oral Ferrous Sulfate
Number analyzed (Participants) | 40 | 39
percentage | 24.30 [19.19 to 29.41] | 8.66 [3.70 to 13.63]
Statistical Analysis 1: Comparison: Ferric Caroboxymaltose vs Oral Ferrous Sulfate; Test type: Superiority; p = 0.0001, ANCOVA; Mean Difference (Final Values) = 15.64

4. Secondary Outcome: Change in Reticulocyte Hemoglobin (Picograms) Content From Baseline to Day 35
Description: Change in reticulocyte hemoglobin (picograms) content from baseline to day 35 was analyzed using a mixed model repeated. The model included terms for the randomization strata (hemoglobin and age categories), baseline ferritin as a reticulocyte hemoglobin content.
Time Frame: Baseline to day 35
Population: Intent to treat
Measure: Least Squares Mean (95% Confidence Interval); unit: picograms
Arm/Group | Ferric Caroboxymaltose | Oral Ferrous Sulfate
Number analyzed (Participants) | 40 | 39
picograms | 6.95 [6.21 to 7.70] | 4.90 [4.15 to 5.65]
Statistical Analysis 1: Comparison: Ferric Caroboxymaltose vs Oral Ferrous Sulfate; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = 2.06

ADVERSE EVENTS:
Time Frame: Day 1 through Day 35
Description: AE will be elicited by nonspecific questions such as "Have you noticed any problems?" Participants will be encouraged to report AEs at their onset. Any AE spontaneously reported by, elicited from the participant, or observed by the physician or study staff, shall be recorded on the appropriate Adverse Event (AE) page of the eCRF. T
Arm/Group | Ferric Caroboxymaltose | Oral Ferrous Sulfate
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT03523117/Prot_003.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT03523117/SAP_001.pdf